CLINICAL TRIAL: NCT04982562
Title: Interest of the 7 Tesla MRI in the Diagnosis of Post-concussion Syndromes Among Patients With Mild Traumatic Brain Injury
Acronym: SPIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPIN
Record Dates: First submitted 2021-06-24; First posted 2021-07-29 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Post-Concussion Syndrome
Keywords: post-concussion Syndrome; diagnosis of 7T MRI in post-concussion syndrom; S100b; mild head trauma
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7T MRI (Other): Seven tesla brain MRI (7T MRI) at day 7 in patients suffering from post concussionnal symptoms after mild traumatic brain injury admitted to emergency departement of Poitiers CHU (University Hospital
  Interventions: Other: 7T MRI

INTERVENTIONS:
Other: 7T MRI — Seven tesla brain MRI (7T MRI) at day 7 in patients suffering from post concussionnal symptoms after mild traumatic brain injury admitted to emergency departement of Poitiers CHU (University Hospital

SUMMARY:
We aimed to conduct a prospective longitudinal interventionnal monocentric study to assess the ability of seven tesla MRI to detect diffuses axonal lesions in patients presenting a post concussional syndrom (PCS) at seven days about a mild traumatic brain injury (MTBI). Our first objective was to evaluate the diagnostic performance of seven tesla MRI runned at seven days after MTBI among patients presenting a PCS.

DETAILED DESCRIPTION:
Among patients admitted in emergency care units in France for mild traumatic brain injury, 10 % will develop post concussionnal symptoms. The variability of the clinical presentation lead to a syndrome at the border of neurology, psychiatry and neuro-traumatology. Ninety per cent of these patients will have a favorable evolution in three to six months while ten per cent will have persistant symptoms : dizziness, headache, nausea, drowsiness, anxio-depressive symptoms, irritability, memory impairments, attentionnal disorders. This conduct to an additionnal medical and social cost (medical re-consultation in emergency services, pharmaceutical expenditure due to over medication, social recognition, deterioration of social and professionnal relationships …). The litterature data show the presence of diffuse axonal lesions (DAL) frequently observed in patients victims of MTBI. These lesions seemed to be correlate with the occurrence of post concussional symptoms. New brain imagery have lead to these discoveries but are not relevant in clinical routine (functionnal MRI, Diffusion Tensor Imaging, tractography). Computed Tomography is often normal and not able to detect these lesions. Standard MRI is not enough sensible for the detection of the DAL. Some autor shows alose that his sensibility decrease in time.

These observations and encouraging results lead us to initiate a prospective interventionnal, longitudinal, pilot study monocentric using seven tesla MRI to evaluate its input in the detection of diffuse axonal lesions among patients presenting post concussionnal symptoms after a mild traumatic brain injury at day seven after they are admitted to our emergency service.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury with glascow included between 13 and 15, with indication of scan
* possibilty of performing an MRI at 7 days
* Patient able to get to MRI at Day 7
* Free consentement to the study
* Any measure of guardianship or curatorship , any link of subordination

Exclusion Criteria:

* Patient does not hospitalized about head trauma
* Inhability to move out for run the seven day MRI
* Contraindication for MRI
* Patient having already consulted the emergency for head trauma requiring imaging
* Patients with psychiatric troubles : bipolarity, panic trouble, depressive trouble, schizophrenia
* Patient already enrolled in the study
* History of brain, tumor or neurosurgery
* Untreated or poorly treated chronic vertigo
* Untreated or poorly treated chronic migraines
* Claustrophobia
* BMI > 40
* Refusal of consent to take part of the study
* No social welfare or inhability to benefit of it by a third party
* Patients with enhanced protection : minor aged under 18 ; person with freedom restriction by justice decision or administrative ; homeliving in health or social establishment ; adult in legal protection
* Pregnant and nursing women

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2024-06-26 (Estimated); Study Completion 2024-06-26 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic performance of 7 Tesla MRI performed of mild head trauma for the occurrence of post-concussion syndrome (PCS) | Day 7
  appearance of diffuse axonal lesions

SECONDARY OUTCOMES:
Evaluate the S100b dosed at admission is correlated with the occurrence of post concussion syndrome after a mild head injury. | Day 0
  Value of S100b dosed at admission
Evaluate the S100b dosed at admission is correlated with diffuse axonal lesion | Day 7, Month 6, Month 12
  appearance of diffuse axonal lesion and S100b dosed at admission
Assess the quality of life of patients suffering for post-cocussion syndrome | Day 7, Month[6;12]
  quality of life EQ-5D-5L questionary (score ranging from levels 1, 2, 3 (without problems) and levels 4,5 (with problems) and GOS-E scales (score ranging from 1.1 (good recovery) to 5 (death).
Correlation the association between the alteration of the anisotropy fraction (AF) and post-concussion syndrome on the MRI diffusion tensor (DTI) sequence | Day 7
  Focal alteration of AF data on a DTI sequence.
Describe the diagnostic performance of the 7 T MRI and quality of life on the occurrence of a post-concussion syndrome | Month [3;6;12]
  Rivermead Post Concussion Scale, ranging from 0 to 4 ; 0 = minimal , 4 = severy problem with 16 items results 64 points maximals (cut-off>12)
Compare the performance obtained on cognitive functioning as a function of cognitive reserve | Month 3
  Attentional Performance : Reaction times, correct, false responses and omissions = percentiles. 5 ≥ pathological. memory disorder : Verbal Learning Test : ≥ -1.65. pathological. bells test. Nb of total omission and a score of Left-Right omission are reported. Pathological > 6 or a left-right score > 2. Visual reproduction . immediate and delayed recall < 7 pathological. Times to name, to read colours. Total errors are also converted in standard notes.Verbal fluencies Nber of words beginning with the letters P,R,S in 1 min. for each letter are summed. The result is z-scored. Perceptual Reasoning index : Block design and Picture Completion. Sum of the standard notes = percentile rank. Verbal Comprehension index : Similarities and Information. Sum of the standard notes = percentile rank. Working Memory index : Arithmetic and Digit Span. Sum of the standard notes = percentile rank.Processing speed index : Code. The standard note = twice to obtain the percentile rank.
Compare in patients the presence of anxio-depressive syndrome | Month 3
  Beck scale (Beck Depression Inventory Scale). The score runs from 0 to 39. 0-3 : no depressed mood; 4-7 : light depressed mood; 8-15 : mild depressed mood; 16 and more : severe depressed mood.
Correlation the association between the presence of a lesion on 7T MRI and the results of various neuropsychological tests. | Month 12
  Attentional Performance : Reaction times, correct, false responses and omissions = percentiles. 5 ≥ pathological. memory disorder : Verbal Learning Test : ≥ -1.65. pathological. bells test. Nb of total omission and a score of Left-Right omission are reported. Pathological > 6 or a left-right score > 2. Visual reproduction . immediate and delayed recall < 7 pathological. Times to name, to read colours. Total errors are also converted in standard notes.Verbal fluencies Nber of words beginning with the letters P,R,S in 1 min. for each letter are summed. The result is z-scored. Perceptual Reasoning index : Block design and Picture Completion. Sum of the standard notes = percentile rank. Verbal Comprehension index : Similarities and Information. Sum of the standard notes = percentile rank. Working Memory index : Arithmetic and Digit Span. Sum of the standard notes = percentile rank.Processing speed index : Code. The standard note = twice to obtain the percentile rank.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France